CLINICAL TRIAL: NCT06703866
Title: Validation of Predictive Model in Value-based Medicine for Lung Cancer and Analysis of Its Implications for Patient Communication
Brief Title: Value-Based Medicine (VBM) for Lung Cancer
Acronym: VBM
Status: Recruiting | Type: Observational
Sponsor: European Institute of Oncology (Other)
Responsible Party: Sponsor
Other Study IDs: IEO 1399
Record Dates: First submitted 2024-03-22; First posted 2024-11-25 (Actual); Last update posted 2024-11-25 (Actual); Status verified 2024-03

CONDITIONS: Lung Cancer
MeSH Terms: conditions — Lung Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Non Small Cell Lung Cancer (NSCLC): Patients with diagnosis of Non Small Cell Lung Cancer (NSCLC) eligible for surgical lung resection (lobectomy/typical and atypical segmentectomy) with or without neo-adjuvant and adjuvant therapy
  Interventions: Other: Non Small Cell Lung Cancer (NSCLC)

INTERVENTIONS:
Other: Non Small Cell Lung Cancer (NSCLC) — Application of "value based medicine" predictive model

SUMMARY:
This is a prospective observational monocentric trial. The primary endpoint is the validation of predictive models. These predictive models will be used to develop a personalized clinical-functional risk profile for estimating in advance, prior to surgery, the probability for a patient to experience surgical complications, pain, fatigue, dyspnea, as well as issues related to physical function, role, social, and emotional well-being, up to 12 months post-discharge.

DETAILED DESCRIPTION:
The goal of this prospective observational monocentric study is to validate a predictive models in patients with diagnosis of non-small cell lung cancer eligible for surgical lung resection (lobectomy/typical and atypical segmentectomy) with or without neo-adjuvant and adjuvant therapy.

Participants will be asked to complete quality of life questionnaires before surgery and then at 30 days, 4 months, 8 months and 12 months post discharge.

The informations collected through questionnaires, along with clinical data will be used to validate the predictive models created.

These models will then be utilized to develop a personalized clinical-functional risk profile for estimating in advance, prior to surgery, the probability for a patient to experience surgical complications, pain, fatigue, dyspnea, as well as issues related to physical function, role, social, and emotional well-being, up to 12 months post-discharge.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 18 years
* Patients with diagnosis of non-small cell lung carcinoma
* Only patients eligible for surgical lung resection (lobectomy/typical and atypical segmentectomy) with or without neo-adjuvant and adjuvant therapy
* Diagnosis of primary non-small cell lung cancer
* Signed Informed Consent
* Patients must be available for follow-up

Exclusion Criteria:

* Patients with benign lesion
* Patients with recurrence who have already undergone lung surgery
* Conditions/pathologies that prevent the ability to give consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with first diagnosis of non-small cell lung carcinoma eligible for surgical lung resection and available for follow up
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2021-01-27 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Creation of a personalized clinical-functional risk profile | 12 months
  Developement of a personalized clinical-functional risk profile for estimating , prior to surgery, the probability for a patient to experience surgical complications, pain, fatigue, dyspnea, as well as issues related to physical function, role, social, and emotional well-being, up to 12 months post-discharge.
  The patient will be asked to complete questionnaires (EORTC QLQ-C30 / EORTC QLQ- LC13) on clinical-functional status and quality of life both before and after surgery, at 30 days, 4 months, 8 months and 12 months after discharge. The information acquired with the questionnaires, together with the clinical information acquired during the healthcare services, will be used to validate and refine the predictive models created and will be used to create a personalized clinical-functional risk profile.

CONTACTS AND LOCATIONS:
Overall Officials: Monica Casiraghi, Principal Investigator — European Institute of Oncology
Locations (1):
- European Institute of Oncology, Milan, Italy